CLINICAL TRIAL: NCT00431990
Title: A Phase I/II Trial of Romidepsin (Depsipeptide) and Bortezomib in Patients With Relapsed Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Celgene Corporation (Industry); Janssen-Cilag Ltd. (Industry)
Responsible Party: Simon Harrison/ Consultant Haematologist, Peter MacCallum Cancer Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06/34
Record Dates: First submitted 2007-02-04; First posted 2007-02-06 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Depsipeptides; romidepsin; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: depsipeptide — Cohort 1. Dose escalation, IV, Weeklyx3 in a 4week cycle. Cohort 2A. 12mg/m2, IV, Weeklyx3 in a 4week cycle. Cohort 2B. 12mg/m2, IV, Weeklyx2 in a 3week cycle.
  Other Names: Romidepsin
Drug: bortezomib — Cohort 1 and 2A. 3.5mg/m2, IV, day 1, 4, 8, 11 in 28 day cycle. Cohort 2B. 3.5mg/m2, IV, day 1, 4, 8, 11 in 21 day cycle
  Other Names: Velcade
Drug: dexamethasone — 20mg for 2 days with each dose of bortezomib

SUMMARY:
The purpose of the first phase of the study is to determine whether, and at what dose, depsipeptide, bortezomib and dexamethasone can be safely administered to patients with Multiple Myeloma. The second phase of the study will establish whether depsipeptide, bortezomib and dexamethasone is effective in the treatment of patients with multiple myeloma. The study will also examine the role of maintenance therapy with depsipeptide.

DETAILED DESCRIPTION:
Several groups have explored the possible synergistic interactions between proteasome and HDAC inhibitors in malignant hematopoietic cells. Bortezomib and HDACIs synergistically induce apoptosis, mitochondrial injury (via BAX), ROS generation and oxidative injury in human leukemia and myeloma cells.

In view of this evidence, we are proposing a trial to examine the clinical effects of combined romidepsin and bortezomib in patients with relapsed/refractory MM. However, there are currently no data as to whether these drugs are safe to administer in combination or at what dose toxicity they may become unacceptable.

Trial Design Open label, single centre, single arm, phase I/II dose escalation trial of bortezomib-dexamethasone with the addition of romidepsin followed by maintenance therapy until disease progression.

Primary objective:

• To determine the maximum tolerated dose (MTD) of romidepsin administered with Bortezomib in patients with relapsed multiple myeloma by the assessment of adverse events and abnormal laboratory values.

Primary endpoint:

• Toxicity evaluation at each of four dose levels presented in the dose-escalation schedule

Secondary objective:

• To determine the efficacy of this combination at the MTD in terms of (i) overall response, (ii) time to progression and (iii) overall survival

Secondary endpoints:

* Overall response (OR), defined as the best response on treatment based on M Protein response criteria with CR documented to EMBT standard and in conjunction with soft tissue plasmacytomas response criteria and corrected serum calcium level.
* Time to progression (TTP), defined as the time from commencement of treatment to the date of first evidence of progressive disease.
* Overall survival (OS), defined as the time from commencement of treatment to the date of death from any cause

ELIGIBILITY:
Inclusion Criteria:

1. Patient was previously diagnosed with multiple myeloma based on standard criteria treated with at least one, but less than 4 lines of therapy, and currently requires further treatment because of relapse from CR or PD.
2. Patient previously treated with bortezomib will be included in the study, if the duration of response was >6mths from the completion of therapy.
3. Patient's age is > 18 yrs
4. Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
5. Patient has given voluntary written informed consent.
6. Female patients of child-bearing potential and male patients with female partners of child-bearing potential, one of whom has not undergone surgical sterilisation must agree to use 2 simultaneous methods of contraception. For female patients, a negative pregnancy test is to be performed within 7 days prior to administration of study drugs.
7. Patient has measurable disease.

   * serum monoclonal protein (SEP) > 5 g/L
   * serum-free light chains (SFLC) > 100 mg/L
   * urine-free light chains (UFLC) > 200 mg/24hr
   * measurable soft tissue (not bone) plasmacytoma (STPC)
8. Patient has a Karnofsky performance status ≥80%.
9. Patient has a life-expectancy >3 months.
10. Patient has the following laboratory values within 14 days before study drug administration:

    * Platelet count ≥50 × 109/L without transfusion support within 7 days
    * Hemoglobin ≥75 g/L without transfusion support within 7 days
    * Absolute neutrophil count (ANC) ≥0.75 × 109/L without the use of growth factors.
    * Corrected serum calcium <14 mg/dL (3.5 mmol/L).
    * Serum potassium ≥ 4.0 mmol/L and serum magnesium ≥ 0.85 mmol/L (electrolytes can be corrected with supplementation. See section 9.7).
    * Aspartate transaminase (AST): ≤2.5 × the upper limit of normal (ULN).
    * Alanine transaminase (ALT): ≤2.5 × the ULN.
    * Total bilirubin: ≤1.5 × the ULN.
    * Calculated or measured creatinine clearance: ≥20 mL/minute.

Exclusion Criteria:

1. Prior severe allergic reactions to bortezomib (Velcade), romidepsin, boron or mannitol
2. Neuropathy > Grade 3 or Neuropathy of Grade 2 with pain > Grade 1 by NCI-CTCAE criteria (v3.0).
3. Patients with the following cardiac risk factors will be excluded from the study (as per the previous NCI trials):

   * Congenital long QT syndrome
   * QTc interval > 480 milliseconds
   * Patients who have had a myocardial infarction within 12 months of study entry.
   * Patients who have active coronary artery disease, e.g. angina as defined by Canadian Class II-IV (Appendix 3).
   * Patients with an ECG showing evidence of cardiac ischemia (ST depression of ≥ 2 mm).
   * Patients with congestive heart failure that meets NYHA Class II to IV definitions (Appendix 4) and/or ejection fraction < 45% by MUGA scan or < 50% by echocardiogram and/or MRI.
   * Patients with a history of sustained VT, VF, Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD).
   * Patients with dilated, hypertrophic, or restrictive cardiomyopathy from prior treatment or other causes (in doubt, see ejection fraction criteria above).
   * Patients with uncontrolled hypertension, i.e. SBP ≥ 160 mm Hg or DBP ≥ 95 mm Hg.
   * Patients with cardiac arrhythmia requiring anti-arrhythmic medication other than beta blocker or calcium channel blocker. Patients in whom digitalis cannot be discontinued are excluded from study.
   * Patients with Mobitz II second degree heart block, that do not have a pacemaker.

   Note: Patients with other cardiac disease may be excluded at the discretion of the principal investigator following consultation with cardiologist.
4. Pregnancy in female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-11; Primary Completion 2011-12 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity | Until progression

SECONDARY OUTCOMES:
Overall response | Until progression
Time to progression | Until progression
Overall survival | Until progression

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Harrison, MBBS, PhD., Principal Investigator — Peter MacCallum Cancer Centre, Australia; Miles Prince, MD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Harrison SJ, Quach H, Link E, Seymour JF, Ritchie DS, Ruell S, Dean J, Januszewicz H, Johnstone R, Neeson P, Dickinson M, Nichols J, Prince HM. A high rate of durable responses with romidepsin, bortezomib, and dexamethasone in relapsed or refractory multiple myeloma. Blood. 2011 Dec 8;118(24):6274-83. doi: 10.1182/blood-2011-03-339879. Epub 2011 Sep 12. PMID 21911830
- See also: Hospital web site — http://www.petermac.org